CLINICAL TRIAL: NCT06644612
Title: A Comparative Study of Light vs Heavy Weighted Polypropylene Mesh in Abdominal Hernia Repair: A Randomized Control Trial Focusing on Surgical Site Infections
Brief Title: Light vs Heavy Weighted Mesh Repair in Primary Abdominal Hernia in Terms of Surgical Site Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: Lady Reading Hospital, Pakistan (Other Government)
Responsible Party: Principal Investigator, Dr Sheraz Fazid, Coordinator in Institute of Public Health and Social Science, Khyber Medical University Peshawar, Khyber Medical University Peshawar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2024/008
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Abdominal Hernia
Keywords: Abdominal Hernia; Surgical Site Infection; Light Weighted Mesh; Heavy Weighted Mesh; Randomized Controlled Trial
MeSH Terms: conditions — Hernia, Abdominal; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated into two groups: one group will undergo hernia repair using light-weighted polypropylene mesh, and the other group will receive heavy-weighted polypropylene mesh. The incidence of SSIs post-operatively will be compared between the two groups.
Who Masked: Participant
Masking Description: Single-blinded trials will be conducted where participants will be unaware of the intervention they will receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group A (Light Mesh Group) (Experimental): All the patients will be administered intravenous Antibiotics two hours before induction of anaesthesia. The surgical site will be shaved if needed after scrubbing the patient. Prolene suture material will be used to anchor the light mesh and suture the skin. A negative pressure drain will be placed if needed. The wound will be dressed with gauze dressing. Post-operatively daily dressing will be done by ward dispenser following full aseptic technique.
  Interventions: Procedure: Light Weight Mesh
- Intervention Group B (Heavy Mesh Group) (Active Comparator): All the patients will be administered intravenous antibiotics two hours before induction of anaesthesia. The surgical site will be shaved if needed after scrubbing the patient.
  Prolene suture material will be used for anchoring the Heavy mesh and for suturing the skin. A negative pressure drain will be placed if needed. The wound will be dressed with a gauze dressing. Post-operatively daily dressing will be done by ward dispenser following full aseptic technique.
  Interventions: Procedure: Heavy Weight Mesh

INTERVENTIONS:
Procedure: Light Weight Mesh — Participants will undergo abdominal hernia repair using light-weighted polypropylene mesh. Standard post-operative care and antibiotic prophylaxis will be provided.
  Arms: Intervention Group A (Light Mesh Group)
Procedure: Heavy Weight Mesh — Participants will undergo abdominal hernia repair using heavy-weighted polypropylene mesh. Standard post-operative care and antibiotic prophylaxis will be provided.
  Arms: Intervention Group B (Heavy Mesh Group)

SUMMARY:
This study compares the incidence of surgical site infections (SSI) in patients undergoing abdominal hernia repair using either light or heavy-weighted polypropylene mesh. The study aims to determine which mesh type results in fewer SSIs, thereby guiding future surgical approaches to abdominal hernia repair.

DETAILED DESCRIPTION:
Hernias, a protrusion of abdominal contents through the abdominal wall, are often treated surgically using synthetic polypropylene mesh. Two varieties of polypropylene mesh exist: light and heavy weighted. The lighter mesh is softer, less allergenic, and potentially leads to fewer post-surgical complications, including SSIs. In contrast, heavier mesh, which has been traditionally used, consists of thicker threads with narrower gaps and has a higher chance of eliciting an immune response. This trial aims to assess the effectiveness of light mesh over heavy mesh in reducing SSIs in abdominal hernia repairs, thereby providing data to support best practices in surgical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15 and above.
* Patients undergoing primary abdominal hernia repair using light or heavy mesh.

Exclusion Criteria:

* Patients with incisional hernias.
* Patients with diabetes mellitus, chronic cough, steroid use, cancer, or immune-compromised status.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) | 10 days
  Incidence of Surgical Site Infection (SSI) within 10 days post-surgery. Using Complete Blood Count (CBC) and site of infection will be checked for the structure affected.

SECONDARY OUTCOMES:
Post-operative Pain | 10 days
  Post-operative pain severity measured using a standardized pain scale (Visual Analogue Scale). Higher scores indicate more severe pain. Scores are interpreted are from 0-4: Mild pain 5-7: Moderate pain, 7-10: Severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Dr Abdul Wahab, Principal Investigator — Lady Reading Hospital, Pakistan
Locations (1):
- Lady Reading Hospital, Pakistan, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interested in the stated study area after its proper monitoring. Data or samples shared will be coded, with no PHI included. Prior permission of the investigators, participants and concerned departments will be obtained.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 12 months after article publication.
Access Criteria: Access can be requested by qualified researchers through proper approval of the investigators.

REFERENCES:
- [Background] Ponten JEH, Leclercq WKG, Lettinga T, Heemskerk J, Konsten JLM, Bouvy ND, Nienhuijs SW. Mesh OR Patch for Hernia on Epigastric and Umbilical Sites (MORPHEUS-Trial): The Complete Two-year Follow-up. Ann Surg. 2019 Jul;270(1):33-37. doi: 10.1097/SLA.0000000000003086. PMID 30339623
- [Background] Rastegarpour A, Cheung M, Vardhan M, Ibrahim MM, Butler CE, Levinson H. Surgical mesh for ventral incisional hernia repairs: Understanding mesh design. Plast Surg (Oakv). 2016 Spring;24(1):41-50. doi: 10.4172/plastic-surgery.1000955. PMID 27054138
- [Background] Eriksen JR, Gogenur I, Rosenberg J. Choice of mesh for laparoscopic ventral hernia repair. Hernia. 2007 Dec;11(6):481-92. doi: 10.1007/s10029-007-0282-8. Epub 2007 Sep 11. PMID 17846703